CLINICAL TRIAL: NCT02863341
Title: Nursing Home Team-Care Deprescribing Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tan Tock Seng Hospital (Other)
Collaborators: Monash University (Other); National Healthcare Group, Singapore (Other Government)
Responsible Party: Principal Investigator, Kua Chong Han, PhD Intern, Tan Tock Seng Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2016/00422
Record Dates: First submitted 2016-07-31; First posted 2016-08-11 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2018-04

CONDITIONS: Fall in Nursing Home; Medication Therapy Management

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (4):
- naive Deprescribing arm (Experimental): Team-based deprescribing practice, Deprescribing Guide
  Interventions: Other: Team-care deprescribing with deprescribing guide
- naive Wait-list Control arm (No Intervention)
- non-naive Deprescribing arm (Experimental): Team-based deprescribing practice, Deprescribing Guide
  Interventions: Other: Team-care deprescribing with deprescribing guide
- non-naive Wait-list Control arm (No Intervention)

INTERVENTIONS:
Other: Team-care deprescribing with deprescribing guide — Beers criteria 2015, STOPP criteria 2014, drug interaction
  Arms: naive Deprescribing arm; non-naive Deprescribing arm

SUMMARY:
This is a multi-centre study in Singapore nursing homes, investigating the factors that affecting deprescribing, and if a team-care based deprescribing standard practice gives superior health and pharmacoeconomic outcomes over current medication review practice.

ELIGIBILITY:
For interview questionnaire:

Inclusion criteria are:

1. Accepted informed consent,
2. The healthcare professional is practicing in the involved nursing homes.

Exclusion criteria are:

1) Decline/unable to provide consent.

For team-care deprescribing study:

Inclusion criteria are:

1. Accepted informed consent (unless cognitive-impaired, with no or un-contactable next-of-kin),
2. Adult aged 65 years and above,
3. Currently on five or more medications.

Exclusion criteria are:

1. Below the age of 65 years of age,
2. Life expectancy of less than 6 months or respite care.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 295 (Actual)
Dates: Start 2016-11; Primary Completion 2018-03 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Fall Risk Assessment Tool (FRAT) score | Change from baseline in FRAT score at 3 months
Change from baseline in Fall Risk Assessment Tool (FRAT) score | Change from baseline in FRAT score at 6 months
Change from baseline in Fall Risk Assessment Tool (FRAT) score | Change from baseline in FRAT score at 12 months
Change from baseline in fall rate | Change from baseline in fall rate at 3 months
Change from baseline in fall rate | Change from baseline in fall rate at 6 months
Change from baseline in fall rate | Change from baseline in fall rate at 12 months

SECONDARY OUTCOMES:
Factors affecting deprescribing | 0 month
  Interview questionnaire
Change from baseline in mean number of medications per subject | Change from baseline in mean number of medications per subject at 3 months
Change from baseline in mean number of medications per subject | Change from baseline in mean number of medications per subject at 6 months
Change from baseline in mean number of medications per subject | Change from baseline in mean number of medications per subject at 12 months
Change from baseline in mean medication cost per subject | Change from baseline in mean medication cost at 3 months
Change from baseline in mean medication cost per subject | Change from baseline in mean medication cost at 6 months
Change from baseline in mean medication cost per subject | Change from baseline in mean medication cost at 12 months
Change from baseline in deprescribing intervention acceptance rate | Change from baseline in deprescribing intervention acceptance rate at 3 months
Change from baseline in deprescribing intervention acceptance rate | Change from baseline in deprescribing intervention acceptance rate at 6 months
Change from baseline in deprescribing intervention acceptance rate | Change from baseline in deprescribing intervention acceptance rate at 12 months
Change from baseline in percentage of drug-related problems (DRPs) | Change from baseline in percentage of DRPs at 3 months
  Medication review form (Hepler/Strand DRP classification system)
Change from baseline in percentage of drug-related problems (DRPs) | Change from baseline in percentage of DRPs at 6 months
  Medication review form (Hepler/Strand DRP classification system)
Change from baseline in percentage of drug-related problems (DRPs) | Change from baseline in percentage of DRPs at 12 months
  Medication review form (Hepler/Strand DRP classification system)

CONTACTS AND LOCATIONS:
Overall Officials: Chong Han Kua, Principal Investigator — Monash University/Tan Tock Seng Hospital
Locations (1):
- Nursing homes, Singapore, Singapore

REFERENCES:
- [Derived] Kua CH, Yeo CYY, Char CWT, Tan CWY, Tan PC, Mak VS, Lee SWH, Leong IY. Nursing home team-care deprescribing study: a stepped-wedge randomised controlled trial protocol. BMJ Open. 2017 May 9;7(5):e015293. doi: 10.1136/bmjopen-2016-015293. PMID 28490560

DOCUMENTS (1):
  • Study Protocol (2017-03-17): https://cdn.clinicaltrials.gov/large-docs/41/NCT02863341/Prot_000.pdf